CLINICAL TRIAL: NCT03038256
Title: Effect of Concurrent Capecitabine-based Long-term Radiotherapy Followed by 4 Cycles XELOX Pre- a Delayed TME Compared With 6 Cycles XELOX post-a Regular Timing TME in Patients With High Risk Rectal Cancer: a Multi-centers, Randomized, Open-Label Trial
Brief Title: Effect of Concurrent Capecitabine-based Long-term Radiotherapy Followed by XELOX Plus TME in Patients With High Risk Rectal Cancer: a Multi-centers, Randomized Controlled, Open-Label Trial
Acronym: EXPLORE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Beijing Friendship Hospital (Other); Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); Shanghai Zhongshan Hospital (Other); Fujian Medical University Union Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Xijing Hospital (Other); Hebei Medical University Fourth Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Affiliated Hospital of Hebei University (Other)
Responsible Party: Principal Investigator, YE Yingjiang, Department of GI Surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12 EXPLORE
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer; Pathological Complete Response; Disease Free Survival
Keywords: High Risk Rectal Cancer; Total neoadjuvant chemoradiotherapy; Lengthening interval between radiotherapy and surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 Cycles XELOX pre- TME (Experimental): experimental group (arm B): concurrent capecitabine-based long-term radiotherapy, 4 cycles of XELOX as neoadjuvant chemotherapy and TME surgery
  Interventions: Drug: concurrent capecitabine-based long-term radiotherapy followed by 4 cycles XELOX and a delayed TME
- 6 Cycles XELOX post- TME (Active Comparator): control group (arm A): concurrent capecitabine-based long-term radiotherapy, TME surgery and 6 cycles of XELOX as adjuvant chemotherapy.
  Interventions: Drug: concurrent capecitabine-based long-term radiotherapy followed by a Regular TME and 6 Cycles XELOX

INTERVENTIONS:
Drug: concurrent capecitabine-based long-term radiotherapy followed by 4 cycles XELOX and a delayed TME — concurrent capecitabine-based long-term radiotherapy: capecitabine 825mg/m2,bid,d1-5, q week with Radiation treatment. Radiation treatment was given at 1·8 Gy per day, 5 days per week for 5-6 weeks, after a 45 Gy radiation dose in 25 fractions to the pelvis, a boost dose of 5·4 Gy in 3 fractions to the tumor bed or concurrent boosted.
  XELOX:
  Oxaliplatin: 130mg/m2,IV,d1; Capecitabine: 1000mg/m2,bid,d1-14; repeated every 3 weeks
  Surgery Procedure:
  Total Mesorectal Excision
  Arms: 4 Cycles XELOX pre- TME
Drug: concurrent capecitabine-based long-term radiotherapy followed by a Regular TME and 6 Cycles XELOX — concurrent capecitabine-based long-term radiotherapy: capecitabine 825mg/m2,bid,d1-5, q week with Radiation treatment. Radiation treatment was given at 1·8 Gy per day, 5 days per week for 5-6 weeks, after a 45 Gy radiation dose in 25 fractions to the pelvis, a boost dose of 5·4 Gy in 3 fractions to the tumor bed or concurrent boosted.
  XELOX:
  Oxaliplatin: 130mg/m2,IV,d1; Capecitabine: 1000mg/m2,bid,d1-14; repeated every 3 weeks
  Surgery Procedure:
  Total Mesorectal Excision
  Arms: 6 Cycles XELOX post- TME

SUMMARY:
The purpose of this study was to evaluate the effect of concurrent capecitabine-based long-term radiotherapy followed by 4 cycles XELOX pre- a delayed TME compared with 6 cycles XELOX post- a Regular Timing TME in patients with high-risk rectal cancer defined by MRI.

DETAILED DESCRIPTION:
This is the randomized controlled, multi-centers, and open-labeled study. Delivering systemic chemotherapy between concurrent capecitabine-based long-term radiotherapy and total mesorectal excision (TME) surgery would be more effectively improved local control rates and improved metastases-free survival rates. The investigators attempted to investigate the effect on pathological response of delivering 4 cycles XELOX between concurrent capecitabine-based long-term radiotherapy and TME with lengthening the interval from radiation to surgery. In this study, the participants with high risk of deeper infiltration, or extramural vessel invasion, or circumferential resection margin involvement, or surrounding organs and structures invaded et al. were recruited. The participants will be randomized (1:1 ratio) to a control and intervention arm. The participants in the control arm will receive best current practice of concurrent capecitabine-based long-term radiotherapy followed by TME and then a 6 cycles of XELOX as standard adjuvant chemotherapy. The participants in the intervention arm will receive concurrent capecitabine-based long-term radiotherapy followed by 4 cycles XELOX as neoadjuvant chemotherapy pre- a delayed TME.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years;
2. Histologically confirmed adenocarcinoma;
3. The rectal adenocarcinoma 0-12cm from the anal margin on Magnetic resonance imaging (MRI) and/or rigid sigmoidoscopy;
4. High risk of rectal cancer defined by high-resolution MRI: tumor invasion 5mm beyond the muscularis propria, or extramural vascular invasion, or circumferential resection margin unsafe, or the lower rectal cancer invades intersphincteric space, or rectal cancer invades the adjacent structures.
5. Eastern Collaborative Oncology Group performance status score of 0 or 2
6. Able and willing to give informed consent to participate.

Exclusion Criteria:

1. Received preoperative chemoradiotherapy for rectal cancer before the recruitment of this study;
2. Have metastatic disease (including non-regional lymph nodes metastases or resectable liver metastases);
3. Other malignancies, non-adenocarcinoma rectal malignancies or rectal malignancies on the basis of inflammatory bowel disease;
4. Emergency surgery due to bowel obstruction, perforation, bleeding, etc.;
5. Abnormality of capecitabine absorption due to gastrointestinal disease e.g. short bowel syndrome, inflammation bowel disease, et al.;
6. Unresectable concurrent intestinal lesions;
7. Concurrent severe infection；
8. Cardiac Disease：uncontrolled or symptomatic cardiac angina，or uncontrolled arrhythmias and hypertension, or severe congestive heart failure grade II or more based on New York Heart Association (NYHA); myocardial infarction within the past 12 months
9. Peripheral neuropathy more than grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE; version 3·0)
10. Bone marrow, liver and kidney function are abnormal e.g., white blood cell ≤ 1.5 × 109 / L; platelet ≤ 100 × 109 / L; Haemoglobin ≤ 80 g/L; Bilirubin > 1.5 times the upper limit; aspartate aminotransferase and alanine aminotransferase > 2.5 times the upper limit; creatinine > 1.5 times the upper limit;
11. Pregnant or lactating women;
12. Life prediction less than 3 months, other severe diseases;
13. Contraindication to MRI; e.g. non-MRI compatible hip prosthesis, cardiac pacemaker;
14. Contraindication to standard chemotherapy including drug interactions and glomerular filtration rate <50 mL/min at baseline;
15. Participators who had been recruited by other clinical trial within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | up to 30days after total mesorectal excision
  Pathological complete response (pCR) rate between control and intervention arm

SECONDARY OUTCOMES:
Disease Free Survival | 3-year
  Disease Free Survival was defined as the time from the date of surgery to the date of the local recurrence, and/or distant disease, or tumor-related death.
R0 of total mesorectal excision rate | up to 30days after total mesorectal excision
  Overall R0 of total mesorectal excision rate between the control and intervention arm
Surgery morbidity | 30 days and 12-months
  Surgical morbidity reported according to Clavien-Dindo classification
quality of surgery | Time of surgery
  Quality of surgery determined using the mesorectal grading system

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Valentini V, van Stiphout RG, Lammering G, Gambacorta MA, Barba MC, Bebenek M, Bonnetain F, Bosset JF, Bujko K, Cionini L, Gerard JP, Rodel C, Sainato A, Sauer R, Minsky BD, Collette L, Lambin P. Nomograms for predicting local recurrence, distant metastases, and overall survival for patients with locally advanced rectal cancer on the basis of European randomized clinical trials. J Clin Oncol. 2011 Aug 10;29(23):3163-72. doi: 10.1200/JCO.2010.33.1595. Epub 2011 Jul 11. PMID 21747092
- [Result] Moran BJ. Predicting the risk and diminishing the consequences of anastomotic leakage after anterior resection for rectal cancer. Acta Chir Iugosl. 2010;57(3):47-50. doi: 10.2298/aci1003047m. PMID 21066983
- [Result] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Result] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Result] Lutz MP, Zalcberg JR, Glynne-Jones R, Ruers T, Ducreux M, Arnold D, Aust D, Brown G, Bujko K, Cunningham C, Evrard S, Folprecht G, Gerard JP, Habr-Gama A, Haustermans K, Holm T, Kuhlmann KF, Lordick F, Mentha G, Moehler M, Nagtegaal ID, Pigazzi A, Pucciarelli S, Roth A, Rutten H, Schmoll HJ, Sorbye H, Van Cutsem E, Weitz J, Otto F. Second St. Gallen European Organisation for Research and Treatment of Cancer Gastrointestinal Cancer Conference: consensus recommendations on controversial issues in the primary treatment of rectal cancer. Eur J Cancer. 2016 Aug;63:11-24. doi: 10.1016/j.ejca.2016.04.010. Epub 2016 May 30. PMID 27254838
- [Result] Chua YJ, Barbachano Y, Cunningham D, Oates JR, Brown G, Wotherspoon A, Tait D, Massey A, Tebbutt NC, Chau I. Neoadjuvant capecitabine and oxaliplatin before chemoradiotherapy and total mesorectal excision in MRI-defined poor-risk rectal cancer: a phase 2 trial. Lancet Oncol. 2010 Mar;11(3):241-8. doi: 10.1016/S1470-2045(09)70381-X. Epub 2010 Jan 25. PMID 20106720
- [Result] Glynne-Jones R, Anyamene N, Moran B, Harrison M. Neoadjuvant chemotherapy in MRI-staged high-risk rectal cancer in addition to or as an alternative to preoperative chemoradiation? Ann Oncol. 2012 Oct;23(10):2517-2526. doi: 10.1093/annonc/mds010. Epub 2012 Feb 23. PMID 22367706
- [Result] Rodel C, Graeven U, Fietkau R, Hohenberger W, Hothorn T, Arnold D, Hofheinz RD, Ghadimi M, Wolff HA, Lang-Welzenbach M, Raab HR, Wittekind C, Strobel P, Staib L, Wilhelm M, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R, Liersch T; German Rectal Cancer Study Group. Oxaliplatin added to fluorouracil-based preoperative chemoradiotherapy and postoperative chemotherapy of locally advanced rectal cancer (the German CAO/ARO/AIO-04 study): final results of the multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Aug;16(8):979-89. doi: 10.1016/S1470-2045(15)00159-X. Epub 2015 Jul 15. PMID 26189067
- [Result] Deng Y, Chi P, Lan P, Wang L, Chen W, Cui L, Chen D, Cao J, Wei H, Peng X, Huang Z, Cai G, Zhao R, Huang Z, Xu L, Zhou H, Wei Y, Zhang H, Zheng J, Huang Y, Zhou Z, Cai Y, Kang L, Huang M, Peng J, Ren D, Wang J. Modified FOLFOX6 With or Without Radiation Versus Fluorouracil and Leucovorin With Radiation in Neoadjuvant Treatment of Locally Advanced Rectal Cancer: Initial Results of the Chinese FOWARC Multicenter, Open-Label, Randomized Three-Arm Phase III Trial. J Clin Oncol. 2016 Sep 20;34(27):3300-7. doi: 10.1200/JCO.2016.66.6198. Epub 2016 Aug 1. PMID 27480145
- [Result] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751